CLINICAL TRIAL: NCT00004148
Title: A Phase I Trial of Intra Lesional RV-B7.1 Vaccine in the Treatment of Malignant Melanoma
Brief Title: Vaccine Therapy in Treating Patients With Unresectable Metastatic Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067380; AECM-99-101; NCI-T99-0006
Record Dates: First submitted 1999-12-10; First posted 2004-02-20 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2006-06

CONDITIONS: Melanoma (Skin)
Keywords: stage III melanoma; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma

ARMS (1):
- Arm I (Experimental): Patients receive rV-B7.1 intralesionally every 4 weeks for 8 weeks (weeks 0, 4, and 8). Treatment continues every 12 weeks in the absence of unacceptable toxicity or disease progression for up to 2 courses. Cohorts of 6-8 patients receive escalating doses of vaccine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 or 3 of 8 patients experience dose limiting toxicities.
  Interventions: Biological: recombinant vaccinia-B7.1 vaccine

INTERVENTIONS:
Biological: recombinant vaccinia-B7.1 vaccine

SUMMARY:
Phase I trial to study the effectiveness of vaccine therapy in treating patients who have unresectable metastatic melanoma. Vaccines may make the body build an immune response to kill tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose of the rV-B7.1 vaccine that elicits a host immune response and is associated with acceptable toxicity in patients with malignant metastatic melanoma.

II. Determine all clinical toxicities associated with this regimen in this patient population.

III. Determine the safety of this regimen in this patient population. IV. Assess evidence of host antimelanoma immune reactivity following this regimen.

V. Determine the effect of this regimen on T-cell immunity. VI. Assess the clinical response in this patient population receiving this regimen.

VII. Evaluate quality of life of these patients during this regimen.

OUTLINE: This is a dose escalation study.

Patients receive rV-B7.1 intralesionally every 4 weeks for 8 weeks (weeks 0, 4, and 8). Treatment continues every 12 weeks in the absence of unacceptable toxicity or disease progression for up to 2 courses. Cohorts of 6-8 patients receive escalating doses of vaccine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 or 3 of 8 patients experience dose limiting toxicities.

Quality of life is assessed before treatment, every 4 weeks, and at end of treatment. Patients are followed every 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven metastatic, unresectable melanoma Dermal, subcutaneous, or lymph node metastases
* Accessible for injection
* Lesions must measure at least 1 cm
* Patients with no prior treatment allowed
* Patients must have one of the following as proof of prior vaccinia immunization:

  * Physician certification
  * Recollection and appropriate vaccination scar site
  * No encephalitis, untreated cerebral metastases, other structural brain lesions, or leptomeningeal disease
  * No ascites or pleural effusions
  * No leukemia or lymphoma

PATIENT CHARACTERISTICS:

* Age: Over 18
* Performance status: ECOG 0-1 Karnofsky 80-100%
* Life expectancy: Greater than 3 months
* WBC greater than 4,000/mm3
* Platelet count greater than 100,000/mm3
* Hemoglobin greater than 10g/dL
* Bilirubin less than 1.5 mg/dL
* Transaminases no greater than 2 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 2 times ULN
* PT/PTT no greater than 2 fold elevation in patients not receiving anticoagulation medications
* No alcoholic cirrhosis
* Creatinine less than 2.0 mg/dL OR creatine clearance greater than 60 mL/min
* No congestive heart failure
* No serious cardiac arrhythmias
* No recent prior myocardial infarction
* No clinical coronary artery disease
* No chronic obstructive pulmonary disease
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No seizure disorders
* No underlying immunosuppressive disorder
* No autoimmune disease HIV negative
* No skin diseases
* No open wounds
* No eczema or other contraindications to vaccinia virus administration
* Patients must be able to avoid high risk individuals (e.g., immunosuppressed patients, children under 3 years, pregnant women, patients with active or a history of eczema, or patients with other skin conditions) for 7-10 days following treatment
* No significant allergy or hypersensitivity to eggs
* No active or chronic infections
* No concurrent medical illness
* No other significant medical disease which would increase risk to patient
* No other prior malignancy within the past 5 years except stage I carcinoma of the cervix or basal cell carcinoma

PRIOR CONCURRENT THERAPY:

* At least 8 weeks since prior immunotherapy and recovered
* No prior live pox virus vector
* No more than 2 prior chemotherapy regimens
* At least 4 weeks since prior chemotherapy and recovered
* At least 4 weeks since prior systemic corticosteroids
* No systemic corticosteroids for concurrent illness
* No concurrent immunosuppressive steroids
* At least 2 weeks since prior radiotherapy and recovered (no bone marrow toxicity)
* At least 6 months since prior radiotherapy for brain metastases and recovered
* At least 4 weeks since prior surgery for management of the primary or metastatic lesions and recovered with remaining measurable disease
* At least 6 months since prior surgery for brain metastases and recovered
* No concurrent immunosuppressive drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 1999-10; Primary Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard L. Kaufman, MD, Study Chair — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein Comprehensive Cancer Center, The Bronx, New York, United States

REFERENCES:
- [Result] Kaufman HL, Deraffele G, Mitcham J, Moroziewicz D, Cohen SM, Hurst-Wicker KS, Cheung K, Lee DS, Divito J, Voulo M, Donovan J, Dolan K, Manson K, Panicali D, Wang E, Horig H, Marincola FM. Targeting the local tumor microenvironment with vaccinia virus expressing B7.1 for the treatment of melanoma. J Clin Invest. 2005 Jul;115(7):1903-12. doi: 10.1172/JCI24624. Epub 2005 Jun 2. PMID 15937544
- [Result] Kaufman HL, Conkright W, Divito J Jr, Horig H, Kaleya R, Lee D, Mani S, Panicali D, Rajdev L, Ravikumar TS, Wise-Campbell S, Surhland MJ. A phase I trial of intra lesional RV-B7.1 vaccine in the treatment of malignant melanoma. Hum Gene Ther. 2000 May 1;11(7):1065-82. doi: 10.1089/10430340050015374. No abstract available. PMID 10811235